CLINICAL TRIAL: NCT05480553
Title: A Phase 3, Placebo-Controlled, Double-Blind Controlled Study of NPC-06 in Patients With Pain Associated With Acute Herpes Zoster
Brief Title: NPC-06 to Pain Associated With Acute Herpes Zoster
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Nobelpharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NPC-06-6
Record Dates: First submitted 2022-07-27; First posted 2022-07-29 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Acute Pain in Herpes Zoster
Keywords: Herpes zoster; fosphenytoin; adjuvant analgesic; acute pain; NPC-06
MeSH Terms: conditions — Herpes Zoster; Acute Pain

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NPC-06 (Experimental)
  Interventions: Drug: NPC-06
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: NPC-06 — 1. Initial dose (Day 1) <Dose> An 18 mg/kg of NPC-06 will be injected by intravenous drip infusion once daily. The maximum dose of the test drug should not exceed 1,200 mg as fosphenytoin sodium.
     <Administration method> Dilute the study drug 3 to 4-fold using physiological saline for intravenous infusion and then administer the solution over 18 minutes.
  2. Maintenance dose(Day 2～7) Maintenance dose on the next day (Day 2) after the initial dose will be mandatory, and will be dosed up to 6 days. Maintenance dose on Day 3 and thereafter will follow the transition criteria for maintenance dose.
  <Dose> A 7.5 mg/kg of NPC-06 will be injected as needed by intravenous drip infusion once daily. The maximum dose of NPC-06 should not exceed 500 mg as fosphenytoin sodium.
  <Administration method> Dilute the study drug 3-to 4-fold using physiological saline for intravenous infusion and then administer the solution over 7 minutes and 30 seconds.
  Arms: NPC-06
Drug: Placebo — 1. Initial dose (Day 1) <Dose> A placebo will be injected by intravenous drip infusion once daily. <Administration method> Dilute the study drug 3 to 4-fold using physiological saline for intravenous infusion and then administer the solution over 18 minutes.
  2. Maintenance dose(Day 2～7) Maintenance dose on the next day (Day 2) after the initial dose will be mandatory, and will be dosed up to 6 days. Maintenance dose on Day 3 and thereafter will follow the transition criteria for maintenance dose.
  <Dose> A placebo will be injected as needed by intravenous drip infusion once daily. Dilute the study drug 3-to 4-fold using physiological saline for intravenous infusion and then administer the solution over 7 minutes and 30 seconds.
  Arms: Placebo

SUMMARY:
To confirm the pain relief effect and the safety of NPC-06 (fosphenytoin sodium hydrate) in patients with pain associated with acute herpes zoster in a placebo-controlled, double-blind, parallel-group, comparative manner.

DETAILED DESCRIPTION:
The eligible patients will be randomized into two groups, and will receive NPC-06 or placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 18 years or older at the time of informed consent.
2. Patients who are male or female.
3. Patients who are inpatient or outpatient.
4. Patients who are diagnosed with herpes zoster and have acute pain.
5. Patients who are within 28 days after the onset of herpes zoster.
6. Patients whose mean NRS pain score is 4 or higher despite the use of the following drugs during the period between 24 hours and 120 minutes before the study drug administration. During this period, one or two of the following drugs should have been used, and the same drug should have been used at least twice.

   * Non-opioid analgesics (excluding its sustained release formulations and topical drugs used for other sites than the target site for efficacy)
   * Ca2＋ channels α2δ ligands (excluding gabapentin)
   * Tramadol (excluding its sustained release formulations)
   * An extract from inflammatory rabbit skin inoculated by vaccinia virus
   * Patients whose NRS pain score immediately before the study drug administration is 4 or higher.

(8) Patients who are able to perform NRS self-assessment appropriately. (9) Patients who gave written informed consent based on their own free will after receiving adequate explanation and fully understanding the details of the explanation in participating in the study.

Exclusion Criteria:

1. Patients who are suspected to be increased intracranial pressure.
2. Patients who are complicated with epilepsy, serious mental or neuropsychiatric disorders (including dementia, Parkinson's disease, or schizophrenia) or consciousness disturbance.
3. Patients who are being treated for malignancy. However, those who do not interfere with daily life and have good general condition may be included in the study.
4. Patients who are being treated for HIV infection or those who are receiving immunosuppressant (including biologics). However, those who do not interfere with daily life and have good general condition may be included in the study.
5. Patients who are being treated for idiopathic trigeminal neuralgia.
6. Patients who have other severe pain that may affect the assessment of pain associated with acute herpes zoster.
7. Patients who have received non-opioid analgesics (excluding its sustained release formulations and topical drugs used for other sites than the target site for efficacy), Ca2＋ channel-α2δ ligands (excluding gabapentin), tramadol (excluding its sustained release formulations), or an extract from inflammatory rabbit skin inoculated by vaccinia virus during the period from 120 minutes before the study drug administration to the start of study drug administration.
8. Patients who have received the following drugs during the period from 24 hours before the study drug administration to immediately before the study drug administration.

   * Non-opioid analgesics (its sustained release formulations)
   * Gabapentin
   * Tramadol (its sustained release formulations)
   * Opioid analgesics
   * Steroidal anti-inflammatory drugs (systemic) for treatment of herpes zoster and pain associated with acute herpes zoster.
   * Antidepressants, antiarrhythmics (excluding those in Vaughan Williams class Ⅱ), NMDA receptor antagonists, centrally acting muscle relaxants, and anesthetics (excluding topical drugs used for other sites than the target site for efficacy).
9. Patients who have sinus bradycardia or advanced conduction disturbance.
10. Patients who have a history of hypersensitivity to hydantoin.
11. Patients who are receiving drugs that are contraindicated in the package insert for fosphenytoin.
12. Patients who have received amenamevir during the period from 24 hours before the study drug administration to immediately before the study drug administration.
13. Patients who are complicated with meningitis or have symptoms of meningeal irritation.
14. Patients who have serious cardiac disease, respiratory disorder, or hepatic or renal dysfunction (as a guide, seriousness corresponding to Grade 3 of "Standards for Classification of Seriousness of Adverse Drug Reactions (Notification No. 80 of the Pharmaceutical Safety Notification ").
15. Patients who are receiving fosphenytoin, phenytoin, ethotoin, or a combination of these drugs or have received these drugs as adjuvant analgesics.
16. Patients who have participated in other clinical study within 3 months of the date of the screening test.
17. Pregnant women, lactating women or patients of childbearing potential during the study period.
18. Patients who are unable to give appropriate contraception in accordance with the instructions of the investigator or sub-investigator (hereafter, the investigators) during the period from after obtaining informed consent to the end of the follow-up period.
19. Other patients who are deemed inappropriate for participation in the study by the investigators.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2022-08-05 (Actual); Primary Completion 2023-05-29 (Actual); Study Completion 2023-08-23 (Actual)

PRIMARY OUTCOMES:
The change of NRS (Numeric Rating Scale:Max10, Min0, higher scores mean a worse outcome) score | 120 minutes after first administration
  Change in the NRS pain score from baseline at 120 minutes after the study drug administration.

CONTACTS AND LOCATIONS:
Locations (20):
- Japan (20):
  - Akemi Dermatology Clinic, Urayasu, Chiba
  - Fukuoka Tokushukai Hospital, Kasuga, Fukuoka
  - Chugoku Rosai Hospital, Kure, Hiroshima
  - Hakodate Central General Hospital, Hakodate, Hokkaido
  - Japanese Red Cross Society Himeji Hospital, Himeji, Hyōgo
  - Koga General Hospital, Koga, Ibaraki
  - Shonan Fujisawa Tokushukai Hospital, Fujisawa, Kanagawa
  - Toyama Dermatologic Clinic, Nichinan, Miyazaki
  - Yoshikawa Skin Clinic, Takatsuki, Osaka
  - Juntendo University Hospital, Bunkyo-ku, Tokyo
  - Sumi Clinic Dermatology Allergology, Meguro City, Tokyo
  - Kurobe City Hospital, Kurobe-shi, Toyama
  - University of Yamanashi Hospital, Chūō, Yamanashi
  - Fukuoka Kinen Hospital, Fukuoka
  - Hakata Pain Clinic, Fukuoka
  - Matsuda Tomoko Dermatological Clinic, Fukuoka
  - National Hospital Organization Kanazawa Medical Center, Kanazawa
  - University Hospital Kyoto Prefectural University of Medicine, Kyoto
  - Kawasaki Medical School General Medical Center, Okayama
  - Shizuoka City Shizuoka Hospital, Shizuoka

IPD SHARING:
Plan to Share IPD: No